CLINICAL TRIAL: NCT00263198
Title: Phase II Study of the Combination of PTK787/ZK222584 and Letrozole in Postmenopausal Women With Advanced Hormone Receptor Positive Breast Cancer
Brief Title: PTK and Letrozole in Post-menopausal Women With Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unacceptable toxicity
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0970
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — vatalanib; Letrozole

ARMS (1):
- Letrozole + PTK787/ZK222584 (Experimental): Letrozole 2.5 mg PO daily for 28 days (patients who have already been treated with letrozole for at least 28 days can skip this part)
  Start cycle 1 with:
  * Letrozole 2.5 mg PO once daily
  * PTK787/ZK222584 250 mg BID PO for 1 week, then 500 mg BID PO for the 2nd week followed by 500 mg qAM and 750 mg QPM PO for the subsequent 2 weeks.
  Subsequent cycles:
  * PTK787/ZK222584 500 mg qAM and 750 mg qPM PO daily
  * Letrozole 2.5 mg PO once daily
  Interventions: Drug: PTK787/ZK222584; Drug: Letrozole

INTERVENTIONS:
Drug: PTK787/ZK222584
Drug: Letrozole

SUMMARY:
The purpose of this study is to test the safety of PTK787/ZK222584 and Letrozole when given in combination, and to see what effects they have on breast cancer that has metastasized.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with metastatic breast cancer, or loco-regional disease recurrence not amenable to treatment by surgery or radiotherapy.
* Postmenopausal status will be defined by any of the following criteria:

  * no spontaneous menses for at least 5 years
  * spontaneous menses within the past 5 years but amenorrheic for at least 12 months and estradiol and/or FSH values in the postmenopausal range (while off aromatase inhibitor therapy; levels can have been taken while on tamoxifen but in this case estradiol should be the parameter assessed)
  * bilateral oophorectomy
  * radiation castration and amenorrheic for at least 3 months
  * the use of an LHRH agonist throughout the duration of the trial (for example goserelin 3.6 mg s.c. monthly)
* Age ≥ 18 years old
* Patients whose tumors are either estrogen-receptor (ER) and/or progesterone-receptor (PgR) positive (10% or more infiltrating cancer cells exhibiting nuclear staining). Patients will be regarded as ER or PgR positive as long as at least one of the tissues assessed was positive. A positive biochemical test is also acceptable.
* Patients must have a WHO Performance Status Grade 0-2
* Newly diagnosed patients who are initiating first line treatment or those patients with known disease who have shown resistance to anti- estrogen therapy (tamoxifen or toremifine).
* Patients currently receiving letrozole or alternative aromatase inhibitors as initial therapy who are without evidence of progressive disease are eligible.
* Patients with bone-only metastasis are eligible.
* Laboratory values ≤ 2 weeks prior to randomization:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L (≥ 1500/mm3)
  * Platelets (PLT) ≥ 100 x 109/L (≥ 100,000/mm3)
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 ULN
  * Serum bilirubin ≤ 1.5 ULN
* Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3.0 x ULN (≤ 5 x ULN if liver metastases present)
* Negative for proteinuria based on dip stick reading OR, if documentation of +1 result for protein on dip stick reading, then total urinary protein

  * 500 mg and measured creatinine clearance (CrCl) ≥ 50 mL/min from a 24- hour urine collection
* Life expectancy ≥ 12 weeks
* Written informed consent obtained according to local guidelines

Exclusion Criteria:

* Patients with tumors which are both estrogen and progesterone receptor negative, or estrogen receptor negative and progesterone receptor unknown or estrogen receptor unknown and progesterone receptor negative
* Patients with a history of adrenalectomy or hypophysectomy
* Patients who developed progressive disease while being treated with an aromatase inhibitor.
* Patients with any of the following:

  * Absolute Neutrophil Count < 1.5 x 109/L
  * Hemoglobin < 9 g/dl
  * Platelet count < 100 x 109/L
  * AST and ALT > 3 times the upper limit of normal or > 5 times the upper limit of normal if liver metastasis are present
  * Bilirubin > 1.5 upper limit of normal
  * Creatinine > 1.5 x upper limit of normal
  * Calcium > 11.6 mg/dL
* History or presence of central nervous system (CNS) disease (i.e., primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis)
* Patients with a history of another primary malignancy ≤ 5 years that has not been treated for curative intent or that the chance of long term remission is judged to be less than 50%.
* Prior chemotherapy <3 weeks prior to registration and/or randomization. Patients must have recovered from all therapy-related toxicities
* Prior biologic or immunotherapy ≤ 2 weeks prior to registration and/or randomization. Patients must have recovered from all therapy-related toxicities
* Patients with a history of treatment with Fulvestrant or Trastuzumab < 6 months prior to registration. Patients must have recovered from all therapy- related toxicities in order to be enrolled.
* Prior full field radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to randomization. Patients must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease
* Major surgery (e.g., laparotomy) ≤ 4 weeks prior to randomization. Minor surgery ≤ 2 weeks prior to randomization. Insertion of a vascular access device is not considered major or minor surgery in this regard. Patients must have recovered from all surgery-related toxicities
* Patients who have received investigational drugs ≤ 4 weeks prior to registration and/or randomization
* Prior therapy with anti-VEGF agents
* Peripheral neuropathy with functional impairment ≥ CTC grade 2 neuropathy, regardless of causality
* Pleural effusion or ascites that causes respiratory compromise (≥ CTC grade 2 dyspnea)
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  * Uncontrolled high blood pressure (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 95 mmHg), history of labile hypertension, or history of poor compliance with an antihypertensive regimen
  * Unstable angina pectoris
  * Symptomatic congestive heart failure
  * Myocardial infarction ≤ 6 months prior to registration and/or randomization
  * Serious uncontrolled cardiac arrhythmia
  * Uncontrolled diabetes (fasting blood sugar > 300 mg/dl)
  * Active or uncontrolled infection
  * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
  * Patients with prolonged QTc > 470 msec on EKG. All patients with a history of congenital or acquired long QTc syndrome.
  * Chronic renal disease
  * Acute or chronic liver disease (e.g., hepatitis, cirrhosis)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK 222584 (i.e., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets)
* Patients with confirmed diagnosis of human immunodeficiency virus (HIV) infection are excluded at the investigator's discretion if it is felt that:

  1) a potential drug interaction between PTK787/ZK 222584 and any of the patient's anti-HIV medications could influence the efficacy of the anti-HIV medication, or 2) it may place the patient at risk due to the pharmacologic activity of PTK787/ZK 222584. Please refer to appendix for a list of examples of substrates of human liver microsomal P450 enzymes
* Patients who are taking therapeutic warfarin sodium (Coumadin) or similar oral anticoagulants that are metabolized by the cytochrome P450 system. Heparin in any formulation is allowed. Please refer to appendix for a list of examples of substrates of human liver microsomal P450 enzymes
* Patients on P450 enzyme inducing anti-epileptics
* Patients who are unwilling or unable to comply with protocol requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-03; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Assess the effect of the combination of letrozole & PTK787/ZK222584 on disease progression. | 24 weeks after starting PTK787/ZK222584

SECONDARY OUTCOMES:
Evaluate the response rate (CR and PR) | Completion of treatment
Evaluate the safety and tolerability of the combination of drugs | 30 days after completion of study treatment
Evaluate the pharmacokinetic profiles of the combination of drugs | Cycle 3 Day 1
Evaluate the modulation of tumor blood flow and blood vessel permeability in response to PTK787/ZK222584 when administered in combination with letrozole using Dynamic Contrast-Enhanced Magnetic Resonance Imaging | Cycle 1 Day 28
Evaluate the effect on circulating tumor cells | Completion of treatment
  Determined by the commerical Immunocon cell search assay
Compare outcome of patients receiving letrozole and PTK787/ZK222584 (cases) with control patients from pivotal trials of letrozole in the first and second line setting. | 30 days after completion of study treatment
  Matching the cases and controls for line of therapy, sites of disease and duration of prior aromatase inhibitor therapy before the study patient initiates PTK787/ZK222584 treatment.
Evaluate polymorphisms in relevant drug metabolism genes to determine the molecular basis for interactions between letrozole and PTK787/ZK222584 should they occur. | Completion of treatment
Correlate serum LDH level with clinical response | Completion of treatment
With additional patient consent, collect peripheral blood cells, serum, plasma, and representative tumor tissue specimens for future correlative science studies | Baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ma, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu